CLINICAL TRIAL: NCT03502369
Title: Randomized, Controlled, Double Blind Trial of Ultrasound Guided Quadratus Lumborum Block for Post Operative Analgesia After Hip Arthroplasty
Brief Title: Ultrasound Guided Quadratus Lumborum Block for Post Operative Analgesia After Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Abdullah Gaber, Registeral, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 050108004
Record Dates: First submitted 2018-04-11; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Adult 90 orthopaedic patient ASA physical status |-||| will be randomly allocated in two groups each one 45 patients, one group will receive the anterior quadratus lumborum block and the other group will not receive the block.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL group (Experimental): Anterior Quadratus lumborum block will be done for all patients of these group. Local anaesthetic (30ml of bupivacaine) will be injected in fascial plane between the quadratus lumborum muscle and Psoas major muscle by using the ultrasound.
  Interventions: Procedure: Anterior Quadratus lamborum block
- C group (No Intervention): Patients of these group will be the control group. The will receive acetaminophen 1g every 8h, ketorolac 30mg ever 12h and as required morphine 2mg for post operative analgesia after hip arthroplasty.

INTERVENTIONS:
Procedure: Anterior Quadratus lamborum block — Local anaesthetic will be injected in the fascial plane between psoas major muscle and quadratus lumborum muscle.
  Other Names: Transmuscular QL block; QL3
  Arms: QL group

SUMMARY:
The study evaluates the effectiveness of anterior quadratus lumborum block for post operative analgesia after hip arthroplasty. Half of the participants will receive ultrasound guided anterior quadratus lumborum block using 30ml bupivacaine 0.375%, while the other half will not receive the block ( control group).

DETAILED DESCRIPTION:
Sensory innervation of the hip region involves branches of the lumbar plexus and sacral plexus. Effective post operative analgesia can be approached by blocking the lumbar plexus at the level of the quadratus lumborum muscle. Quadratus lumborum block has several approach methods (anterior, lateral, posterior, and intramuscular). Anterior quadratus lumborum block also known as transmuscular QL block or QL3, the local anaesthetic (30ml of bupivacaine 0.375%) is injected between the psoas major muscle (PM) and the quadratus lumborum muscle (QL). Therefore, the anterior quadratus lumborum block may generate analgesia from T10 to L4 covering the sensory innervation of the hip region.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status |-||| , scheduled to undergo unilateral hip replacement via lateral approach.

Exclusion Criteria:

* patient refusal.
* History of neurological/neuromuscular, psychiatric, dementia preventing proper comprehension.
* coagulation disorders.
* History of allergy to the study medication.
* Infection overlying the injection site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity assessment | every hour for the first 4 post operative hours and then every 4 hours for the rest of the 24 post operative hours.
  Patients will be trained to use visual analogue scale which consists of 10cm line, 0 cm equivalent to no pain and 10 cm denoting the worst imaginable pain.

SECONDARY OUTCOMES:
Total amount of post operative morphine (mg). | any time in the first 24 post operative hours.
  Total amount of post operative morphine (mg) used as rescue analgesia and the first time of its request.

OTHER OUTCOMES:
Patient satisfaction. | every hour in the first 4 post operative hours and then every 4 hours for the rest of the 24 post operative hours.
  Patient satisfaction with pain control will be assessed on a four point scale 1.Excellent 2.Good 3.fair 4.poor

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.

REFERENCES:
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Result] Sauter AR, Ullensvang K, Niemi G, Lorentzen HT, Bendtsen TF, Borglum J, Pripp AH, Romundstad L. The Shamrock lumbar plexus block: A dose-finding study. Eur J Anaesthesiol. 2015 Nov;32(11):764-70. doi: 10.1097/EJA.0000000000000265. PMID 26426575